CLINICAL TRIAL: NCT01746342
Title: A Randomized, Controlled, Clinical Trial of Continuous Positive Airway Pressure Treatment of Obstructive Sleep Apnea-Hypopnea in Multiple Sclerosis
Brief Title: Sleep Apnea in Multiple Sclerosis Positive Airway Pressure Trial
Acronym: SAMSPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Multiple Sclerosis Society of Canada (Primary funding agency) (Unknown); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Philips Respironics (Industry); VitalAire Incorporated (Respiratory Therapist time) (Unknown)
Responsible Party: Principal Investigator, Dr John Kimoff, Co-Principal Investigator: with Dr Daria Trojan, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSSC-G004
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea-hypopnea in Multiple Sclerosis Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Effective CPAP (Active Comparator): Continuous positive airway pressure: effective fixed level determined by polysomnographic titration
  Interventions: Device: Effective continuous positive airway pressure (CPAP)
- Sham CPAP (Sham Comparator): Continuous positive airway pressure device modified by manufacturer to deliver minimal pressure
  Interventions: Device: Sham continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Effective continuous positive airway pressure (CPAP)
  Arms: Effective CPAP
Device: Sham continuous positive airway pressure (CPAP)
  Arms: Sham CPAP

SUMMARY:
Fatigue is highly prevalent among multiple sclerosis (MS) patients and has pervasive adverse effects on daily functioning and quality of life. The investigators found in a recent study that obstructive sleep apnea-hypopnea (OSAH) is the most common sleep abnormality in multiple sclerosis (MS) patients. There was also a significant relationship between OSAH and higher fatigue scores in MS patients. Preliminary work from the investigators in this group of subjects shows that treatment of sleep disorders (mostly OSAH) can improve fatigue and other symptoms in some MS patients. However, it is now necessary to systemically test the effect of OSAH treatment in a randomized, controlled study, to be sure that it really does improve fatigue and other symptoms. The best treatment for OSAH in the general population is continuous positive airway pressure (CPAP). This treatment has been well tolerated by most MS patients who have used the device at the investigators' center. This project will therefore be a randomized, controlled, clinical trial of CPAP in MS patients with OSAH. The effects of six months of CPAP treatment on fatigue as well as sleep quality, somnolence, pain, disability, and quality of life will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis by a neurologist based on standard criteria (Annals Neurol 2011; 69:292-302)
* Expanded Disability Status Scale score of 0 to 7.0
* MS-relapse free for >30 days prior to screening
* Pittsburgh sleep quality Index > 5
* Fatigue Severity Scale score >=4
* Montreal Cognitive Assessment (MoCA) >= 26
* diagnosis of OSAH by polysomnography showing AHI >= 15 events/h of sleep
* forced vital capacity >60% predicted

Exclusion Criteria:

* pregnancy or planned pregnancy
* psychiatric conditions which could preclude compliance with informed consent, study procedures, or study requirements
* other significant neurological, pulmonary, otorhinological, and medical disorders
* major depression within the past year
* any value of >1.5 times the upper limit or <0.75 the lower limit of the reference range for any standard clinical hemogram and biochemistry determinations which is clinically significant
* current treatment for OSAH
* presence of another untreated sleep disorder which is clinically significant
* very severe OSAH (safety criterion)defined as an AHI >30 with either a 4% O2 desaturation index >15 events/h OR work in a safety-critical position OR an ESS score >=15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-02; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Six months

SECONDARY OUTCOMES:
Fatigue Scale for Motor and Cognitive Functions | Three & Six months
Epworth Sleepiness Scale | Three & Six months
Pittsburgh Sleep Quality Index | Three & Six months
Pain visual analog scale | Three & Six months
Multiple Sclerosis-specific quality of life measure-54 (MSQOL-54) | Three & Six months
Fatigue Severity Scale | Three months
  Primary outcome measure is FSS at six months
Expanded Disability Status Scale | Three & Six months
  Standard scale for evaluation of Multiple Sclerosis-related disease disability
Center for Epidemiological Studies-Depression Scale | Three & Six months
Cognitive evaluation | Six months
  Montreal Cognitive Assessment (MoCA) and Tower of London-Drexel University
Polysomnographic variables | Six months
  Standard complete polysomnographic measures of sleep and respiration
Objective CPAP compliance | Three and Six Months
  Standard measures of CPAP use and efficacy from machine microprocessor

CONTACTS AND LOCATIONS:
Overall Officials: John Kimoff, MD, Principal Investigator — McGill University; Daria Trojan, MD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Khadadah S, Kimoff RJ, Duquette P, Jobin V, Lapierre Y, Benedetti A, Johara FT, Robinson A, Roger E, Bar-Or A, Leonard G, Kaminska M, Trojan DA. Effect of continuous positive airway pressure treatment of obstructive sleep apnea-hypopnea in multiple sclerosis: A randomized, double-blind, placebo-controlled trial (SAMS-PAP study). Mult Scler. 2022 Jan;28(1):82-92. doi: 10.1177/13524585211010390. Epub 2021 Apr 23. PMID 33890515